CLINICAL TRIAL: NCT04581213
Title: Effect of Anesthesia Induction on Cerebral Hemodynamic in Children
Acronym: PEDICACHE
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Florent BAUDIN, Principal Investigator, St. Justine's Hospital
Other Study IDs: 2020_2747
Record Dates: First submitted 2020-09-16; First posted 2020-10-09 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Anesthesia; Reaction; Children, Only
Keywords: General anesthesia; Children
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: General anesthesia — Children under general anesthesia for an elective surgery, aged between 6 months and 5 years old, ASA 1-2.

SUMMARY:
General anesthesia induces hemodynamic changes, notably a reduction of arterial blood pressure going up to 30%, that may impact cerebral perfusion and oxygenation.The purpose of this study is to assess the impact of anesthesia on the cerebral oxygenation, the perfusion of the brain (assessed with transcranial doppler), and the depth of anesthesia in children between 6 months and 5 years old during the induction of general anesthesia (induced with sevoflurane and/or IV agents). It is expected that the cerebral hemodynamic will be maintained despite systemic variations.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia for elective surgery
* American Society of Anesthesiologists score 1 and 2
* Written informed consent obtained from the parents or legal tutors.

Exclusion Criteria:

* 3 unsuccessful attempts of IV access
* ultrasound device non available
* neurologic comorbidity

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under general anesthesia for an elective surgery, aged between 6 months and 5 years old, ASA 1-2.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Changes in NIRS values during induction | baseline and 1 minute after intubation
  Changes in cerebral Near infra-red spectrometry values
Changes in cerebral velocity of the middle cerebral artery during induction | baseline and 1 minute after intubation
Changes of Response Entropy (RE) value during induction | baseline and 1 minute after intubation
Changes of State Entropy (SE) value during induction | baseline and 1 minute after intubation
  Depth of anesthesia

SECONDARY OUTCOMES:
Changes in NIRS values after induction | At 1 minute, 3 minutes after intubation and at the start of surgery
Change in cerebral velocity of the middle cerebral artery after induction | At 1 minute, 3 minutes after intubation and at the start of surgery
Changes of arterial blood pressure during induction | At baseline and 1 minute after intubation
Changes of Response Entropy (RE) values after induction | At 1 minute, 3 minutes after intubation and at the start of surgery
Endtidal Co2 after induction | 1 minute after intubation
Changes of State Entropy (SE) value after induction | At 1 minute, 3 minutes after intubation and at the start of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte Justine Hospital, Montreal, Quebec, Canada